CLINICAL TRIAL: NCT03623815
Title: A Functional Magnetic Resonance Imaging Investigation Into the Effects of Transcranial Direct Current Stimulation on Information Processing in Healthy Volunteers
Brief Title: A Functional Magnetic Resonance Imaging Investigation of Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MS-IDREC-C2-2015-003
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Placebo controlled crossover design
Who Masked: Outcomes Assessor
Masking Description: Double blinding was carried out using a blinding code randomly assigned to each participant by a separate party. This code was entered into the transcranial direct current stimulation device by the investigator to deliver the stimulation. The investigator was not unblinded until initial analysis was complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tDCS followed by active tDCS (Other): Within subjects design. This group received sham (placebo) transcranial direct current stimulation (tDCS) for 20 minutes in session one. At least one month later this group received 2mA of active tDCS for 20 minutes in session two.
  Interventions: Other: transcranial direct current stimulation
- Active tDCS followed by sham tDCS (Other): Within subjects design. This group received 2mA of active transcranial direct current stimulation (tDCS) for 20 minutes in session one. At least one month later this group received sham (placebo) tDCS for 20 minutes in session two.
  Interventions: Other: transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulatory technique that uses weak electrical current to increase (with anodal) or decrease (with cathodal) the probability of brain activity in the stimulated region. This typically has acute effects relating to cortical activity levels which last up to one hour.
  This intervention delivers 20 minutes of 2mA bipolar balanced tDCS, with anodal tDCS delivered to the left dorsolateral prefrontal cortex (DLPFC) and simultaneously cathodal tDCS delivered to the right DLPFC. In the sham condition 40 seconds of stimulation is delivered.
  Other Names: tDCS

SUMMARY:
This study evaluates the effect of frontal cortex transcranial direct current stimulation (tDCS) on the neural correlates of threat processing in healthy volunteers with a high level of trait anxiety. All participants received both active and sham tDCS and underwent a functional imaging scan whilst carrying out an attentional control task with fearful distractors.

DETAILED DESCRIPTION:
There is a growing body of evidence suggesting that repeated administration of prefrontal transcranial direct current stimulation (tDCS) is a potential effective treatment for depression through restoring a left/right imbalance in frontal brain activity (Boggio et al., 2008; Loo et al., 2012) and improving top down control of anxiety responses.

An initial exploratory study was carried out in 2012 (Ironside et al 2015) to examine the effects of tDCS on emotional processing in healthy volunteers using a range of tasks and questionnaires. Using a dot probe task, which measures attention to happy or fearful faces, it was found that tDCS has the potential ability to reverse an attentional bias to fearful faces seen in the placebo group. This indicates that anxiety responses may be modified using tDCS and therefore this follow on study seeks to further explore the role of tDCS in trait anxiety and investigate the neural correlates of this with fMRI.

The present study uses behavioural and neuroimaging results to examine how tDCS affects emotional processing relevant to trait anxiety. A within-subjects design increases the power of the study, given limited resources to carry out extensive neuroimaging. Our working hypothesis is that tDCS may alter activity in cortical regions relevant to attentional control and anxiety.

The findings of this study will be used to determine parameters for future patient studies, involving participants with generalized anxiety disorder or major depression. The ultimate aim, explored through further studies, is to understand and improve how tDCS might be used in the treatment of these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Healthy female adults, right handed, aged 18-45 years.
* Participants will be asked to fill in a pre-screening online anxiety questionnaire (STAI-T) and will be invited to participate in the study if they score high within the normal range on trait anxiety.

Exclusion Criteria:

* Any current significant medical condition.
* Any current or past psychological disorder (for example depression or anorexia).
* Any family history of extreme mood fluctuations (such as elated mood states)
* Any current medications (except for contraceptive treatment) or herbal remedies such as St John's wort.
* Any current pregnancy or likelihood of becoming pregnant during the study.
* Any participation in any other psychological or medical experiment involving taking any kind of drugs, within the last 3 months.
* Previous participation in a brain stimulation study will be taken into account and advice will be sought from the secondary supervisor on whether they should be included, based on the type of stimulation received, the location of the stimulation and the number of sessions. If the secondary supervisor advises that the nature of the stimulation previously received could affect the results of this study, the participant will not be included.
* Participants should not be claustrophobic, have a heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.
* Any other contraindication to magnetic resonance imaging or transcranial current stimulation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2015-10-06 (Actual)

PRIMARY OUTCOMES:
The change in neural activity during an attentional control task after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  A comparison of neural activity (blood oxygenation level dependent response) during an attentional control task after real versus sham tDCS.

SECONDARY OUTCOMES:
The change in accuracy in an attentional control task after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  A comparison of behavioural test results (accuracy in attentional control task) after real versus sham tDCS.
The change in reaction time in an attentional control task after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  A comparison of behavioural test results (mean reaction time in milliseconds in attentional control task) after real versus sham tDCS.
The change in self report anxiety after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  Differences in anxiety symptoms after sham versus real tDCS will be quantified by the change in self report anxiety scores (State-Trait Anxiety Inventory (STAI)) after sham tDCS and real tDCS.
The change in sadness/happiness after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  Differences in sadness/happiness after sham versus real tDCS will be quantified by the change in self report visual analogue scale with sad at 0 and happy at 100 after sham tDCS and real tDCS.
The change in hostility/friendliness after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  Differences in hostility/friendliness after sham versus real tDCS will be quantified by the change in self report visual analogue scale with hostile at 0 and friendly at 100 after sham tDCS and real tDCS.
The change in calmness/tenseness after sham versus real tDCS | Outcome measure quantifies the change between measurement taken after real tDCS versus sham tDCS (order counterbalanced). The time period from the first measurement to the second and final measurement is no less than 30 days and no more than 60 days.
  Differences in calmness/tenseness after sham versus real tDCS will be quantified by the change in self report visual analogue scale with calm at 0 and tense at 100 after sham tDCS and real tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Harmer, PhD, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loo CK, Alonzo A, Martin D, Mitchell PB, Galvez V, Sachdev P. Transcranial direct current stimulation for depression: 3-week, randomised, sham-controlled trial. Br J Psychiatry. 2012 Jan;200(1):52-9. doi: 10.1192/bjp.bp.111.097634. PMID 22215866
- [Background] Boggio PS, Zaghi S, Fregni F. Modulation of emotions associated with images of human pain using anodal transcranial direct current stimulation (tDCS). Neuropsychologia. 2009 Jan;47(1):212-7. doi: 10.1016/j.neuropsychologia.2008.07.022. Epub 2008 Aug 3. PMID 18725237
- [Background] Ironside M, O'Shea J, Cowen PJ, Harmer CJ. Frontal Cortex Stimulation Reduces Vigilance to Threat: Implications for the Treatment of Depression and Anxiety. Biol Psychiatry. 2016 May 15;79(10):823-830. doi: 10.1016/j.biopsych.2015.06.012. Epub 2015 Jun 17. PMID 26210058